CLINICAL TRIAL: NCT06402279
Title: The Effectiveness of Early Hemoperfusion in Patients With Extremely Severe COVID-19 After Intubation on a Ventilator
Brief Title: Hemoperfusion Efferon СT for the Extremely Severe Form of COVID-19
Status: Completed | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-ct-2020-02
Record Dates: First submitted 2024-05-05; First posted 2024-05-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19; mesoporous styrene-divinylbenzene copolymer; cytokines adsorption; hemoperfusion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basic therapy + Efferon CT: Patients in group 1 (n = 65) received basic COVID-19 medication: 2 to 5 days before hemosorption, they all received anti-inflammatory drugs, glucocorticoid therapy (16 to 24 mg/day of dexamethasone), oxygen therapy, and heparin. The transfer to an intensive care unit (ICU) was accompanied by transfer to a non-invasive ventilator.
  Interventions: Device: Efferon CT therapy
- Baseline therapy: Group 2 patients (n=65) were matched to patients of group 1 and received basic COVID-19 drug therapy and no hemoperfusion procedure using Efferon CT device.

INTERVENTIONS:
Device: Efferon CT therapy — Efferon CT is a cylindrical body made of polycarbonate, filled with spherical granules of polymer hemocompatible macroporous styrene-divinylbenzene copolymer of super cross- linked type and isotonic sodium chloride solution. The device is manufactured according to TU 32.50.50-001-12264678-2018, has passed the necessary tests and is registered in Russia as a medical product RZN 2019/8886. Hemoperfusion procedures were performed using the Efferon CT device no later than 6 hours after the start of invasive ventilation. Hemosorption was performed twice within 12 hours, with an interval of 24 hours between hemoperfusion.
  Groups: Basic therapy + Efferon CT

SUMMARY:
The development of acute respiratory and renal failure of COVID-19 patients is associated with an excessive immune response and hyperproduction of anti-inflammatory cytokines, which leads to impaired endothelial function and a dysregulated balance between the coagulation and fibrinolytic systems in the blood. These factors contribute to the development of multi-organ failure, sepsis, and high mortality rates.In the absence of effective etiotropic therapy for COVID-19, it is necessary to search for alternative, pathogenetically based treatment approaches, including extracorporeal methods of homeostasis support. This observational study examines the effect of early hemoperfusion using the Efferon CT device for the treatment of patients with severe forms of COVID-19 after their intubation on a ventilator.

DETAILED DESCRIPTION:
On March 11, 2020, the World Health Organization (WHO) declared COVID-19 a global pandemic. This disease is characterized by a variety of symptoms, many of which can lead to multiple organ failures and critical conditions.Timely removal of cytokines and other medium-molecular substances from the body using sorption techniques can not only help restore the balance between pro-inflammatory and anti-inflammatory mediators, but also in some clinical situations, prevent the deterioration of vital organ function or create conditions that allow for the reversal of multiple organ dysfunction.The accumulated experience of using various devices for sorption of low- and medium-molecular toxins creates a pathophysiological basis for the development of effective methods for the use of extracorporeal hemoperfusion in the treatment of the most severe forms of COVID-19.

This study examines the effects of early hemoperfusion, using the Efferon CT device, for the treatment of severe cases of COVID-19 in patients after intubation on a ventilator.

Efferon CT (Efferon JSC, Moscow, Russia) is a device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by removing excess cytokines, myoglobin, endogenous and exogenous toxic substances from the patient's blood. The device is manufactured according to TU 32.50.50-001-12264678-2018, passed the necessary tests and is registered in Russia as a medical device RZN 2019/8886.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extremely severe COVID-19 no later than 6 hours after the start of intubation on a ventilator
* Patients over 18 years and under 72 years old

Exclusion Criteria:

* Pregnancy or the first 3 months after childbirth
* Clinical or laboratory findings of sepsis
* Acute bleeding
* Presense of cancer in anamnesis
* Surgical interventions
* Acute kidney injury (KDIGO > I)
* Charlson comorbidity index > 5
* Thrombocytopenia with a platelet count less than 100x109/L
* Patients in the first 6 months after acute cerebrovascular accident or acute myocardial infarction
* Patients who have previously undergone extracorporeal detoxication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes, over 18 years and under 72 years old with extremely severe COVID-19 after the start of mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Effect of Efferon CT hemoperfusion on Ventilator-free days (VFDs) | 1-60 days
  VFDs is a composite outcome measure that combines survival and duration of ventilation.

SECONDARY OUTCOMES:
Effect of Efferon CT hemoperfusion on SOFA scores | 1-10 days
  Value of indicators on the Sequential Organ Failure Assessment (SOFA) Score. Each organ system received a score ranging from 0 (normal) to 4 (most abnormal), with a minimum SOFA score of 0 and a maximum SOFA score of 24.
Effect of Efferon CT hemoperfusion on pulmonary oxygen metabolism function | 1-10 days
  Value of oxygenation index (PaO2 / FiO2).
Effect of Efferon CT hemoperfusion on KDIGO stage | 1-10 days
  Degree of acute renal injury.
Effect of Efferon CT hemoperfusion on the need for norepinephrine | 1-10 days
  The number of people who require continuous administration of norepinephrine

CONTACTS AND LOCATIONS:
Overall Officials: Yakovlev Alexey, PhD,MD, Principal Investigator — Nizhny Novgorod regional clinical hospital named after N.A.Semashko
Locations (1):
- Alexey Yakovlev, Nizhny Novgorod, Russia

REFERENCES:
- [Background] Yakovlev AY, Ilyin YV, Bershadsky FF, Selivanov DD, Pevnev AA, Trikole AI, Popov AY, Pisarev VM. Efficacy of hemoadsorption in the severe course of COVID-19. Front Med (Lausanne). 2025 Mar 6;12:1491137. doi: 10.3389/fmed.2025.1491137. eCollection 2025. PMID 40115785